CLINICAL TRIAL: NCT03097627
Title: Intravenous Indocyanine Green for Localization of Intra-thoracic Lesions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yolonda Colson, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015P002271
Record Dates: First submitted 2017-03-13; First posted 2017-03-31 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple
Keywords: Indocyanine Green; Near-infrared imaging
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules | interventions — Indocyanine Green

STUDY DESIGN:
Masking Description: There is no masking in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ICG Intervention (Experimental): The intervention to be administered is intravenous indocyanine green for intra-thoracic lesion localization and use of a near infrared camera to detect the ICG. All study subjects will receive this same intervention; there is only one arm.
  Interventions: Drug: ICG Intervention; Device: Near Infrared Camera

INTERVENTIONS:
Drug: ICG Intervention — The intervention to be administered is the drug indocyanine green.
  Other Names: Indocyanine Green
Device: Near Infrared Camera — The intervention to detect the administered drug, indocyanine green.

SUMMARY:
This is a clinical trial to evaluate the intravenous administration of indocyanine green (ICG) as a method of intra-thoracic lesion localization. The primary purpose is to determine if intravenous ICG allows us to identify intra-thoracic lesions.

DETAILED DESCRIPTION:
* This study is designed to determine the safety and feasibility of intra-operative localization of thoracic lesions following intravenous injection of indocyanine green (ICG), determine if intravenous ICG leads to the intra-operative detection of intra-thoracic lesions or metastatic lymph nodes not readily identifiable on conventional diagnostic imaging modalities, and determine if intravenous ICG improves surgical resection.
* At the time of surgery, the indocyanine dye will be injected intravenously. The investigators will use a dose of 0.5 mg/kg administered prior to VATS.
* The "filtered" near-infrared light causes the indocyanine green dye to fluoresce so that the surgeon can identify the lesions most likely to contain tumor cells.The surgeon will also look at lymph nodes to see if metastatic disease can be found in this location using this technique. The lymph nodes are processed to look for metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intra-thoracic lesions that require resection for therapeutic or diagnostic purposes as recommended by their thoracic surgeon.
* 18 years of age or older
* Documented, signed, dated informed consent obtained prior to any study specific procedures being performed

Exclusion Criteria:

* Subjects who do not wish to have subsequent surgical resection
* A medical condition such as uncontrolled infection or cardiac disease that, in the opinion of the treating surgeon, makes resection unreasonably hazardous for the patient
* Pre-operative spirometry that suggests the patient is at high risk or cannot undergo resection of the primary tumor.
* Iodide or seafood allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and feasibility) of intra-operative localization of thoracic lesions following intravenous injection of indocyanine green (ICG) | 5 years
  In this initial proof-of-concept pilot trial for patients undergoing surgical resection of suspicious intra-thoracic lesions, the investigators will demonstrate that IV ICG is a safe and feasible method for lesion localization. The investigators will demonstrate this across a variety of intra-thoracic pathology including primary lung cancer, pulmonary metastases, mesothelioma, mediastinal tumors, and potentially infectious sources such as aspergilloma. The investigators will measure safety based on number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Determine if intravenous ICG leads to the intra-operative detection of intra-thoracic lesions or metastatic lymph nodes not readily identifiable on conventional diagnostic imaging modalities | 5 years
  The investigators will determine if lesions can be identified that were not seen on pre-operative imaging either because they were too small, missed, or ill-defined. In addition, many lesions such as vague ground glass opacities, which could represent scarring or a slow growing bronchoalveolar cancer, may be targeted with IV ICG, and thus aiding in the decision to resect a given lesion. Lymph nodes that contain disease may also uptake IV ICG. If a lymphadenectomy is indicated for standard of care, NIR positive nodes will be noted.
Determine if intravenous ICG improves surgical resection | 5 years
  In cases of malignancy, performing an adequate oncologic resection (i.e. negative margins) or debulking is crucial to the prognosis of a patient with an intra-thoracic malignancy. Simultaneously, a surgeon must minimize the amount of resected healthy tissue to preserve lung function. Therefore, the investigators will assess the histologic status of the margin in all patients in which the lesion was ICG positive. The investigators will also maintain records of patients undergoing IV ICG to obtain intra-operative characteristics (i.e. successful lesion localization) and long-term events (i.e. local recurrence).

CONTACTS AND LOCATIONS:
Overall Officials: Yolonda Colson, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to share any individual participant data with other researchers.